CLINICAL TRIAL: NCT06938009
Title: Pediatric Resuscitation Neuroprognostication and Outcomes Registry
Brief Title: Dutch Registry of Pediatric Cardiac Arrest
Acronym: PROGNOSE
Status: Recruiting | Type: Observational
Sponsor: Matthijs de Hoog (Other)
Collaborators: Amsterdam UMC (Other); Radboud University Medical Center (Other); University Medical Center Groningen (Other); Maastricht University Medical Center (Other); UMC Utrecht (Other); Zoll Medical Corporation (Industry); Stichting Vermeer14 (Unknown); Leiden University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Matthijs de Hoog, Prof. dr., Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: MEC-2023-0133
Record Dates: First submitted 2025-04-07; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Arrest (CA); Pediatric ALL
Keywords: Pediatric cardiac arrest; Neuroprognostication; Long-term outcomes; Observational registry
MeSH Terms: conditions — Heart Arrest; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric cardiac arrest patient: The study cohort consists of pediatric patients under the age of 18 who have experienced a cardiac arrest-either in-hospital (IHCA) or out-of-hospital (OHCA)-in the Netherlands. Eligible patients must have received care from emergency medical services (EMS) or been admitted to one of the seven participating academic pediatric hospitals following the arrest.
  Cardiac arrest is defined as the absence of a palpable pulse or the need for chest compressions lasting at least one minute, in line with European Resuscitation Council guidelines. Both basic life support (BLS) and advanced pediatric life support (APLS) protocols apply.

SUMMARY:
The goal of this observational study is to understand the long-term outcomes of children in the Netherlands who experience cardiac arrest, either in or outside of the hospital. The main questions it aims to answer are:

What are the survival rates and neurological outcomes in children after cardiac arrest?

What types of emergency and post-resuscitation care are provided, and how do they impact long-term recovery?

How do children and their families function over time after the event?

Researchers will analyze data from routine medical records and follow patients through standard outpatient visits. No extra procedures will be required beyond normal care. For those who survive to hospital discharge, additional follow-up data will be collected with consent.

Participants will:

Be children under 18 years old who have had a cardiac arrest and were treated in one of the seven participating academic hospitals

Have their routine medical care data collected anonymously

Be invited (if surviving) for follow-up visits at 3, 12, and 24 months post-arrest and at specific ages (5, 8, 12, and 17 years) to assess physical and psychological recovery

DETAILED DESCRIPTION:
The PROGNOSE study (Pediatric Resuscitation Neuroprognostication and Outcomes Registry) is a prospective, multicenter, observational patient registry established to improve understanding of short- and long-term outcomes following pediatric cardiac arrest (CA) in the Netherlands. The study focuses on both out-of-hospital (OHCA) and in-hospital cardiac arrest (IHCA) in children under 18 years of age.

Given the rarity yet severity of pediatric CA, the registry aims to collect a large dataset to identify patterns in care, outcomes, and recovery trajectories to ultimately improve treatment strategies and prognosis. The study is considered non-WMO (not subject to the Dutch Medical Research Involving Human Subjects Act), as it involves no additional interventions beyond standard clinical care.

Registry Objectives and Scope The primary objective is to evaluate diagnostic practices and long-term functional and neuropsychological outcomes in pediatric patients post-cardiac arrest. Key secondary objectives include determining the incidence and etiology of pediatric CA in the Netherlands, analyzing survival to discharge, and characterizing post-Return of Circulation (ROC) care.

Data will be collected longitudinally during standard outpatient follow-up visits at specified intervals (3, 12, and 24 months post-arrest; and at the ages of 5, 8, 12, and 17 years, depending on the age at CA event). No study-specific interventions will be performed.

Data Collection and Source Verification

All data collected in this registry will be sourced from routine clinical care and medical records from seven Dutch academic (pediatric) hospitals. Data will be abstracted from:

Emergency services records

Inpatient hospital and ICU documentation

Follow-up outpatient clinic assessments

Neuropsychological and functional evaluations using validated tools (e.g., PCPC, POPC, FSS)

The data will be pseudo-anonymized using unique study IDs. Only site-specific investigators will have access to the link between study ID and patient identity.

Quality Assurance and Monitoring

A robust quality assurance framework has been put in place to ensure data integrity, including:

Data validation procedures: Data entries will be checked against predefined rules for logic, consistency, and range validation in the electronic data capture (EDC) system (Castor EDC).

Source data verification (SDV): Periodic audits by local site PIs will compare registry entries against source data (e.g., EHRs) for completeness and accuracy.

Site monitoring: The coordinating center (Erasmus MC) will provide oversight and perform routine cross-site reviews to ensure harmonized data collection.

Data dictionary: A detailed data dictionary defines all collected variables, including their source, coding schemes (e.g., ICD, MedDRA where applicable), and interpretation ranges.

Standard Operating Procedures (SOPs)

Standard operating procedures have been established to guide the entire registry lifecycle, including:

Site initiation and training

Patient screening and enrollment processes

Data entry and validation procedures

Procedures for obtaining (delayed) informed consent at follow-up

Change management and version control of registry forms

Procedures for data sharing and publication

Statistical Analysis Plan Given its quality improvement nature, no formal sample size calculation was performed. Instead, the registry aims to enroll all eligible pediatric CA cases nationwide, allowing the creation of a comprehensive, hypothesis-generating dataset.

Descriptive statistics will summarize demographics, event characteristics, interventions, and outcomes.

Longitudinal analysis of neuropsychological function and functional status will be performed using repeated-measures ANOVA or mixed-effects modeling.

Comparative statistics (e.g., logistic regression) will be used to identify predictors of survival and favorable neurological outcome. Covariates will be selected based on literature and tested for collinearity. Multivariate models will report odds ratios with 95% confidence intervals.

Missing data will be addressed using appropriate imputation techniques, depending on the mechanism of missingness (e.g., multiple imputation for random missing data).

Plan for Missing Data

To manage incomplete records and potential attrition in follow-up:

All missing values will be coded according to reason (e.g., not applicable, patient deceased, declined follow-up).

Patterns of missingness will be explored. If data are missing at random, multiple imputation may be used in analysis.

Data collection tools prompt required fields and flag missing values to reduce omissions during entry.

Informed Consent and Ethics Due to the emergent nature of CA and the high mortality rate, an exception from consent procedure is employed for initial data collection. For survivors, informed consent is sought at follow-up outpatient visits, as part of standard care. Data are de-identified and used solely for research purposes. No images or human materials are collected.

The study complies with the General Data Protection Regulation (GDPR), the Dutch "Code Goed Gedrag," and the Declaration of Helsinki.

Data Storage and Access Pseudo-anonymized data are stored securely in Castor EDC, managed by Erasmus MC.

Each center has access only to its own data.

A Data Transfer Agreement (DTA) governs anonymized data sharing for multicenter publications.

Data will not be shared outside the EU.

No end date is set for the registry; it will remain open for ongoing data entry and hypothesis generation.

Dissemination Plan Findings from the registry will be disseminated through peer-reviewed publications, with a goal of generating multicenter analyses and contributing to national and international guideline development. A first multicenter manuscript is expected within approximately five years from the start of the registry.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients under the age of 18
* Experienced in-hospital or out-of-hospital cardiac arrest in the Netherlands
* Attended by emergency medical services or admitted to one of the seven participating Dutch academic pediatric hospitals
* Cardiac arrest defined as absence of palpable pulse or need for chest compressions lasting ≥1 minute
* Arrest managed under European Resuscitation Council guidelines (BLS/APLS)

Exclusion Criteria:

* Cardiac arrest occurring in neonates younger than 24 hours of age
* Cardiac arrest occurring in a neonatal intensive care unit (NICU) setting

Ages: 24 Hours to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients under 18 years of age who experienced a cardiac arrest, either in-hospital or out-of-hospital, in the Netherlands. Eligible patients must have received chest compressions for at least one minute and been treated by emergency medical services or admitted to one of seven participating Dutch academic pediatric hospitals. Neonates under 24 hours old and NICU arrests are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Long-term Neurological Outcome (PCPC) | At 3, 12, and 24 months post-cardiac arrest; and at ages 8, 12, and 17 years, depending on age at event
  Neurological outcome will be assessed using the Pediatric Cerebral Performance Category (PCPC) scale, a validated functional outcome measure ranging from 1 to 6. A score of 1 indicates normal age-appropriate cerebral performance, while higher scores reflect increasing levels of neurological impairment: mild (2), moderate (3), severe (4), coma or vegetative state (5), and death (6). Lower scores indicate better neurological function. The highest available follow-up score will be used as the primary neurological outcome measure.
Long-term Neurological Outcome (POPC) | At 3, 12, and 24 months post-cardiac arrest; and at ages 8, 12, and 17 years, depending on age at event
  Overall functional outcome will be assessed using the Pediatric Overall Performance Category (POPC) scale, a validated tool measuring global functional status in children following critical illness or injury. Scores range from 1 (normal) to 6 (death), with higher scores indicating greater overall disability. POPC complements the PCPC by evaluating broader aspects of daily functioning.
Long-term Neurological Outcome (FSS) | At 3, 12, and 24 months post-cardiac arrest; and at ages 8, 12, and 17 years, depending on age at event
  Functional outcome will also be measured using the Functional Status Scale (FSS), a detailed, domain-specific assessment covering six areas: mental status, sensory, communication, motor function, feeding, and respiratory status. Each domain is scored from 1 (normal) to 5 (very severe dysfunction), with a total score ranging from 6 to 30. Lower total scores indicate better overall function.
Neuropsychological Functioning in Pediatric Survivors (composite IQ) | At 12 and 24 months after cardiac arrest
  Neuropsychological outcomes will be assessed using standardized, age-appropriate cognitive and behavioral tests administered during follow-up. The assessment includes:
  Wechsler Intelligence Scale for Children (WISC-V) or Bayley Scales of Infant Development (Bayley-III) depending on age: Composite IQ or developmental index (range varies by age, mean = 100, SD = 15).
  Unit of Measure:
  Standardized test scores (mean ± SD) and proportion of patients with clinically significant impairment (%)
Neuropsychological Functioning in Pediatric Survivors (BRIEF-2 or BRIEF-P) | At 12 and 24 months after cardiac arrest
  Neuropsychological outcomes will be assessed using standardized, age-appropriate cognitive and behavioral tests administered during follow-up. The assessment includes:
  Behavior Rating Inventory of Executive Function (BRIEF-2 or BRIEF-P): T-scores, where higher scores indicate more executive dysfunction (mean = 50, SD = 10).
  Unit of Measure:
  Standardized test scores (mean ± SD) and proportion of patients with clinically significant impairment (%)
Neuropsychological Functioning in Pediatric Survivors (CBCL) | At 12 and 24 months after cardiac arrest
  Neuropsychological outcomes will be assessed using standardized, age-appropriate cognitive and behavioral tests administered during follow-up. The assessment includes:
  Child Behavior Checklist (CBCL): Total problem score, higher scores indicate more behavioral/emotional problems (T-score, mean = 50, SD = 10).
  Unit of Measure:
  Standardized test scores (mean ± SD) and proportion of patients with clinically significant impairment (%)
Neuropsychological Functioning in Pediatric Survivors (PedsQL) | At 12 and 24 months after cardiac arrest
  Neuropsychological outcomes will be assessed using standardized, age-appropriate cognitive and behavioral tests administered during follow-up. The assessment includes:
  Pediatric Quality of Life Inventory (PedsQL): Total score from 0 to 100; higher scores reflect better quality of life.
  Unit of Measure:
  Standardized test scores (mean ± SD) and proportion of patients with clinically significant impairment (%)

SECONDARY OUTCOMES:
Incidence and Cause of Cardiac Arrest | At the time of in-hospital or out-of-hospital cardiac arrest, during initial hospital evaluation
  Differentiated by IHCA and OHCA
  First documented rhythm and suspected etiology
Pre-hospital Interventions Performed (Composite) | At time of cardiac arrest event, as documented during emergency response and initial hospital admission
  This is a composite outcome measure indicating whether any of the following pre-hospital interventions were performed during the cardiac arrest event:
  Bystander-performed basic life support (BLS)
  Use of an automated external defibrillator (AED)
  Initiation of extracorporeal cardiopulmonary resuscitation (ECPR)
  The presence of any one or more of these interventions will qualify as a positive occurrence for the composite measure.
  Unit of Measure:
  Proportion of patients (%) who received at least one of the listed interventions.
  Presentation:
  All components of the composite measure will be presented together in a single summary table.
Duration of Cardiopulmonary Resuscitation (CPR) | At the time of the cardiac arrest event, as documented during emergency medical response and initial hospital admission.
  The total duration, in minutes, of cardiopulmonary resuscitation performed during the cardiac arrest event. This includes both basic and advanced life support provided by bystanders and emergency medical services prior to return of spontaneous circulation or termination of resuscitation efforts.Unit of Measure:
  Minutes
Return of Circulation (ROC) | Time Frame: During initial hospital admission following cardiac arrest
  Whether return of spontaneous circulation was achieved following cardiac arrest, as documented by clinical and physiological parameters. Unit of Measure: Proportion of patients (%)
Survival to Hospital Discharge | Time Frame: During initial hospital admission following cardiac arrest
  Whether the patient survived until discharge from the initial hospital admission following cardiac arrest. Unit of Measure: Proportion of patients (%)
In-Hospital Mortality | During initial hospital admission following cardiac arrest
  Death during initial hospital admission following cardiac arrest. If applicable and available, the presumed or documented cause of death will also be recorded. Unit of Measure: Proportion of patients (%)
Brain Magnetic Resonance Imaging (MRI) Findings | During initial hospital admission following cardiac arrest. Within 7 days after cardiac arrest.
  Brain MRI will be assessed within 7 days after cardiac arrest to evaluate the presence and extent of hypoxic-ischemic brain injury. Findings will be categorized as no injury, focal injury, or extensive injury based on predefined scoring of cortex/white matter and deep gray matter involvement. Unit of measure: Proportion of patients (%) with each MRI injury category (no injury, focal, or extensive injury).
Electroencephalography (EEG) Background Assessment | At 24 hours after return of circulation following cardiac arrest.
  EEG recordings obtained 24 hours after cardiac arrest will be assessed both quantitatively and visually. Quantitative EEG (qEEG) features-such as amplitude and continuity-will be extracted and used to predict 12-month survival. Visual classification will follow standardized critical care EEG terminology, categorizing background as continuous with normal amplitude or other patterns. Unit of measure: Proportion of patients (%) per EEG background category (e.g., continuous ≥20 μV, burst suppression, isoelectric)
Blood Biomarker Analysis | Within the first 72 hours after cardiac arrest
  Blood biomarkers associated with neurological injury and outcome will be measured during the early post-resuscitation phase. Examples may include neuron-specific enolase (NSE), S100 calcium-binding protein B (S100B), and other relevant markers. Values will be used to support neuroprognostication and correlated with long-term outcome. Unit of Measure: Concentration (e.g., ng/mL) and proportion of patients with elevated levels (%)
Family/Caregiver Outcomes PedsQL-FIM | At 3, 12, and 24 months after the cardiac arrest event
  Parent and family well-being will be assessed using validated questionnaires at multiple time points during follow-up. Instruments include:
  Pediatric Quality of Life Family Impact Module (PedsQL-FIM): Total score ranges from 0 to 100; higher scores indicate better functioning.
  Unit of Measure:
  Mean score per questionnaire (with standard deviation) and proportion of parents with clinically relevant distress (%)
Family/Caregiver Outcomes HADS | At 3, 12, and 24 months after the cardiac arrest event
  Parent and family well-being will be assessed using validated questionnaires at multiple time points during follow-up. Instruments include:
  Hospital Anxiety and Depression Scale (HADS): Subscale scores for anxiety and depression each range from 0 to 21; higher scores indicate greater symptom burden.
  Unit of Measure:
  Mean score per questionnaire (with standard deviation) and proportion of parents with clinically relevant distress (%)

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Buysse, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (7):
- Netherlands (7):
  - Radboud umc, Nijmegen, Gelderland
  - MUMC, Maastricht, Limburg
  - Amsterdam UMC, Amsterdam, North Holland
  - UMCG, Groningen, Provincie Groningen
  - LUMC, Leiden, South Holland
  - Erasmus MC, Rotterdam, South Holland
  - UMCU, Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results reported in publications from the PROGNOSE registry will be shared. This includes de-identified clinical data and outcome measures, along with the data dictionary and statistical analysis plan. IPD will be shared to support transparency and enable reproducibility of analyses described in the protocol paper.
Supporting Information: Study Protocol, SAP
Time Frame: IPD and supporting documents will become available upon publication of the protocol paper.
Access Criteria: Access to IPD will be available through the published protocol paper. Researchers may request additional clarification or documentation by contacting the study team. Use of data must be for scientific, non-commercial purposes, and in accordance with ethical and privacy standards.

REFERENCES:
- [Derived] Albrecht M, Hunfeld M, Arkesteijn-Muit A, Dulfer K, de Hoog M, de Jong G, de Jonge R, Lamore A, Nadkarni V, Buysse C; PROGNOSE Group Collaborative Investigators. A Dutch nationwide pediatric cardiac arrest registry with long-term follow-up - towards an international prognostication guideline. Resusc Plus. 2025 May 9;24:100976. doi: 10.1016/j.resplu.2025.100976. eCollection 2025 Jul. PMID 40491775